CLINICAL TRIAL: NCT04510779
Title: Monitoring Heart Failure Patients Using Heart Rate Variability Measured by the Apple Watch
Brief Title: Apple Watch Heart Failure Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AppleWatch
Record Dates: First submitted 2020-08-10; First posted 2020-08-12 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Heart Failure Patients (Experimental): This will be a single arm study of heart failure patients with acute decompensation
  Interventions: Device: Apple Watch

INTERVENTIONS:
Device: Apple Watch — Apple Watch is a smartwatch developed by Apple Inc. The heart rate variability function will be used.

SUMMARY:
This is a pilot/feasibility study on the accuracy of HRV as measured by the Apple Watch on heart failure patients who are admitted to the hospital with heart failure exacerbation. The primary aim is to observe a statistically significant improvement in the HRV of acutely decompensated heart failure patients upon discharge when compared to admission, implying the utility of HRV measured by Apple Watch as a monitor for cardiovascular health.

DETAILED DESCRIPTION:
Heart failure (HF) is a complex clinical syndrome. It is caused by structural or functional impairments, which interfere with the ability of heart muscles to fill or eject blood. The prevalence of HF exceeds 7 million in the United States alone.(1) Despite improving survival, HF hospitalization rates has remained stable, which reflects persisting difficulties in managing existing disease. (2) Specifically, readmission rates may be as high as 50% by 6 months after an admission for HF management. (2) Caring for HF patients exceeds 30 billion annually and is largely driven by hospitalizations.2 Innovative, at-home surveillance tools are needed to reduce hospital admissions and to drive down the overall societal burden of this disease. (3)

HF is characterized by periodic exacerbations due to volume overload and fluid congestion that impairs perfusion to the organs.(2) Accurate assessment of volume status is, therefore, key for early detection of impending exacerbation. Currently, there is no single, objective method of assessment, relying on a combination of tools including physical examination, weight, pulmonary artery catheter or echocardiography.(4) However, these measures are subjective, invasive, or impractical for monitoring patients at home. Unique body habitus and comorbidities of individual patient further complicates assessment of volume status.(4) The future of heart failure management, therefore, lies in the development of a telemonitoring system that is convenient to use and accessible for patients at home, while quantitatively understanding individual characteristics.(4)

Cardiovascular health is closely related to the imbalances of the autonomic nervous system.(5) Heart rate variability (HRV), the degree of fluctuation in the interval between consecutive heartbeats, has been recognized as a reliable marker of autonomic activity.(5) HRV has been shown to be depressed in patients with congestive heart failure (CHF) and to correlate with disease severity. (6) Furthermore, abnormal HRV parameters are independently associated with incident CHF in asymptomatic, older adults. (7)

HRV is conventionally measured using a 24-hour Holter monitor, which is sensitive, but inconvenient and impractical for home monitoring.(5) Newer studies have shown not only the reliability of short term (5-minute) or ultra-short term (<5 minute) analysis of electrocardiographic recordings, but also that of wearable monitors amenable for use at home.(9-11) In particular, HRV parameters measured by Apple Watch (Cupertino, California) were shown to agree with those measured by a validated chest best heart rate monitor.(12)

The usefulness of the study is to validate the utility of wearable heart monitors such as the Apple Watch in accurately measuring heart rate variability, a dynamic marker of cardiovascular health, and correlating it with the health status specifically of heart failure patients. Validating this will allow wearable monitors to record HRV remotely from home, facilitating telemonitoring and preventing hospitalizations.

ELIGIBILITY:
Inclusion Criteria:

* Age > or = 22
* Patients admitted to Tufts Medical Center for acute decompensated heart failure
* Left ventricular ejection fraction greater than 35%
* Able to consent

Exclusion Criteria:

* Pacemaker rhythm
* Arrhythmia, e.g. atrial fibrillation, atrial flutter, frequent ectopic beats
* prior history of heart transplant or ventricular assist device
* pregnant

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Difference of Standard Deviation of NN Intervals upon Discharge Compared to Admission | 1-2 Weeks
  Standard Deviation of NN Intervals is a time domain heart rate variability parameter. The value upon discharge after medical management should be statistically greater compared to admission value.

CONTACTS AND LOCATIONS:
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roger VL. Epidemiology of heart failure. Circ Res. 2013 Aug 30;113(6):646-59. doi: 10.1161/CIRCRESAHA.113.300268. PMID 23989710
- [Background] Desai AS. Home monitoring heart failure care does not improve patient outcomes: looking beyond telephone-based disease management. Circulation. 2012 Feb 14;125(6):828-36. doi: 10.1161/CIRCULATIONAHA.111.031179. No abstract available. PMID 22331920
- [Background] Murray CM, Agha SA, Rathi S, Germany RE. The evaluation and monitoring of volume status in congestive heart failure. Congest Heart Fail. 2008 May-Jun;14(3):135-40. doi: 10.1111/j.1751-7133.2008.05640.x. PMID 18550924
- [Background] Heart rate variability. Standards of measurement, physiological interpretation, and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Eur Heart J. 1996 Mar;17(3):354-81. No abstract available. PMID 8737210
- [Background] Musialik-Lydka A, Sredniawa B, Pasyk S. Heart rate variability in heart failure. Kardiol Pol. 2003 Jan;58(1):10-6. PMID 14502297
- [Background] Patel VN, Pierce BR, Bodapati RK, Brown DL, Ives DG, Stein PK. Association of Holter-Derived Heart Rate Variability Parameters With the Development of Congestive Heart Failure in the Cardiovascular Health Study. JACC Heart Fail. 2017 Jun;5(6):423-431. doi: 10.1016/j.jchf.2016.12.015. Epub 2017 Apr 5. PMID 28396041
- [Background] Ferrario M, Moissl U, Garzotto F, Cruz DN, Clementi A, Brendolan A, Tetta C, Gatti E, Signorini MG, Cerutti S, Ronco C. Effects of fluid overload on heart rate variability in chronic kidney disease patients on hemodialysis. BMC Nephrol. 2014 Feb 4;15:26. doi: 10.1186/1471-2369-15-26. PMID 24490775
- [Background] Nussinovitch U, Elishkevitz KP, Katz K, Nussinovitch M, Segev S, Volovitz B, Nussinovitch N. Reliability of Ultra-Short ECG Indices for Heart Rate Variability. Ann Noninvasive Electrocardiol. 2011 Apr;16(2):117-22. doi: 10.1111/j.1542-474X.2011.00417.x. PMID 21496161
- [Background] Karp E, Shiyovich A, Zahger D, Gilutz H, Grosbard A, Katz A. Ultra-short-term heart rate variability for early risk stratification following acute ST-elevation myocardial infarction. Cardiology. 2009;114(4):275-83. doi: 10.1159/000235568. Epub 2009 Aug 18. PMID 19690410
- [Background] Hernando D, Roca S, Sancho J, Alesanco A, Bailon R. Validation of the Apple Watch for Heart Rate Variability Measurements during Relax and Mental Stress in Healthy Subjects. Sensors (Basel). 2018 Aug 10;18(8):2619. doi: 10.3390/s18082619. PMID 30103376
- [Background] Tanindi A, Olgun H, Celik B, Boyaci B. Heart rate variability in patients hospitalized for decompensated diastolic heart failure at admission and after clinical stabilization. Future Cardiol. 2012 May;8(3):473-82. doi: 10.2217/fca.12.24. PMID 22642636